CLINICAL TRIAL: NCT00559481
Title: Effect of Oral Ketoconazole on the Pharmacokinetics of Oral Dexamethasone and Oral Hydrocortisone in Patients With Androgen Independent Prostate Cancer
Brief Title: Ketoconazole, Dexamethasone, and Hydrocortisone in Treating Patients With Prostate Cancer That Did Not Respond to Androgen-Deprivation Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: I 93506; RPCI-I-93506
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; Ketoconazole; Hydrocortisone

INTERVENTIONS:
Drug: dexamethasone
Drug: ketoconazole
Drug: therapeutic hydrocortisone
Procedure: pharmacological study

SUMMARY:
RATIONALE: Studying samples of blood in the laboratory from patients with cancer receiving ketoconazole together with dexamethasone and hydrocortisone may help doctors learn more about how these drugs are used by the body.

PURPOSE: This randomized clinical trial is studying how ketoconazole, dexamethasone, and hydrocortisone act in the body of patients with prostate cancer that did not respond to androgen-deprivation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the pharmacokinetics of oral dexamethasone with and without oral ketoconazole in patients with androgen-independent prostate cancer.
* To compare the pharmacokinetics of oral hydrocortisone with and without oral ketoconazole in these patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral dexamethasone twice daily on days 1-14, oral ketoconazole 3 times daily on days 2-14 and 30-42, and oral hydrocortisone twice daily on days 29-42.
* Arm II: Patients receive oral hydrocortisone twice daily on days 1-14, oral ketoconazole 3 times daily on days 2-14 and 30-42, and oral dexamethasone twice daily on days 29-42.

In both arms, patients may receive ketoconazole and hydrocortisone as standard salvage therapy off study.

In both arms, patients undergo blood sample collection on days 1, 14, 29, and 42 for pharmacokinetic studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of prostate cancer
* Must have failed standard androgen-deprivation therapy

  * Evidence of rising PSA

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Creatinine ≤ 2.0 mg/dL
* AST and ALT < 4 times upper limit of normal
* Bilirubin < 2.0 mg/dL
* No active congestive heart failure
* No allergy to ketoconazole, dexamethasone, hydrocortisone, or to one of the components of dexamethasone, hydrocortisone, or ketoconazole
* No active infection
* No uncontrolled glaucoma
* No active peptic ulcer disease
* No uncontrolled diabetes mellitus
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy

PRIOR CONCURRENT THERAPY:

* More than 2 weeks since prior and no concurrent drugs known to interact with study treatment

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of oral dexamethasone with and without oral ketoconazole
Pharmacokinetics of oral hydrocortisone with and without oral ketoconazole

CONTACTS AND LOCATIONS:
Overall Officials: Donald L. Trump, MD, Principal Investigator — Roswell Park Cancer Institute